CLINICAL TRIAL: NCT05622994
Title: Efectos de un Antagonista/Agonista Inverso Del Receptor CB1 (Rimonabant) Sobre la Capacidad Para la deambulación en Lesionados Medulares Incompletos
Brief Title: Effects of CB1 Antagonist/Reverse Agonist Rimonabant on Walking Abilities in Incomplete Spinal Cord Injury
Acronym: RIMOFATSCI-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Principal Investigator, Antonio Oliviero, Antonio Oliviero, Hospital Nacional de Parapléjicos de Toledo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHNP-CT003
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries
Keywords: walking abilities; Rimonabant; Endurance; Incomplete SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rimonabant

STUDY DESIGN:
Intervention Model Description: Placebo controlled parallel design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rimonabant (Active Comparator): Rimonabant 5mg
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Rimonabant

INTERVENTIONS:
Drug: Rimonabant — Rimonabant 5mg per day is administered for 90 days. The comparator is placebo for the same duration.
  Other Names: Placebo

SUMMARY:
This is a placebo controlled study comparing Rimonabant 5 mg per day for 90 days with placebo for the same period. Objective is to improve walking abilities of spinal cord injury individuals (incomplete lesions) and demonstrate that it is a safe treatment in spinal cord injury population.

DETAILED DESCRIPTION:
This is a placebo controlled study comparing Rimonabant 5 mg per day for 90 days with placebo for the same period.

Main goal are to test safety and efficacy (impairment of walking abilities teste with the 6 min walking test) of Rimonabant in a specific population (incomplete spinal cord injury).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 yo and <75yo
* Non progressive spinal cord injury
* Incomplete lesion (AIS C or D)
* Neurological level between C4 and L1
* Chronic stage (>1 year since injury)
* Preserved walking ability for at least 5 m (aid allowed)
* Capability to provide informed consent
* For fertile women, possibility to use anti conceptive methods

Exclusion Criteria:

* Age <18 yo or >75
* AIS A, B or E
* Neurological level above C4 or below L1
* Subacute stage (<1 year since injury)
* Preserved walking ability for less than 5 m (aid allowed)
* Pregnancy or breast feeding
* For fertile women, impossibility to use anti conceptive methods
* anticoagulant treatment
* Hypothyroidism
* Severe bone, kidney or liver disfunction
* Impossibility to reach the hospital
* Impossibility to rovide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Safety) | 120 days
  Number of AE
Biochemical and urine analysis (safety) | 120 days
  Number of participants with clinically significant abnormal laboratory tests results
ECG (safety) | 120 days
  Number of participants with clinically significant abnormal ECG readings
Hospital Anxiety and Depression Scale (HAD) (safety | 120 days
  Range 0-21(higher values more severe)
Modified Ashworth Scale (safety) | 90 days
  Range 0-4 (higher values more severe)
Penn Scale (safety) | 90 days
  Range 0-4 (higher values more severe)
Pain numeric rating scale (safety) | 90 days
  Range 0-10 (higher values more severe)
Questionnaire of falls (safety) | 120 days
  Number of falls
6 min walking test (efficacy) | 90 days
  6 min walking test (meters and number of stops are reported)

SECONDARY OUTCOMES:
10 m test (efficacy) | 90 days
  Time to walk 10 m (no stops are allowed)
Borg Scale (efficacy) | 90 days
  Borg Scale punctuation after 6 min waking test. Range 0-10.
Motor Score (efficacy) | 90 days
  Motor Score (ISNCSCI). Range 0-20 (higher values less severe)
Fatigue Severity Scale (FSS) (Efficacy) | 90 days
  FSS puntuación. Range 0-7 (higher values more severe)
Patient global impression of changes (PGIC) (efficacy) | 90 days
  PGIG score. Range 1-7 (higher values indicate worsening)
European Quality of Life -5 Dimensions (EQ-5D) (efficacy) | 90 days
  EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 3 problem levels corresponding to patient response choices (higher values worst). A quality-of-life score is obtained according to the answers to the questionnaires (algorithm to calculate the score in euroqol.org). The maximum score is 1 that indicates excellent quality of life (range for Spanish version 0.5-1).
Health state visual analogically scale (efficacy) | 90 days
  Range 0-100 mm (higher values indicate higher health state )
Spinal Cord Independence Measures, SCIM (efficacy) | 90 days
  Range 0-100 (higher values indicate higher independence )

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Oliviero, MD, PhD, Principal Investigator — Hospital Nacional de Parapléjicos
Locations (1):
- Hospital Nacional de Paraplejicos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No